CLINICAL TRIAL: NCT05676411
Title: Efficacy of Combination of Topical Benzoyl Peroxide and Electrocautery Skin Incision in Eradicating Cutibacterium Acnes From Surgical Wounds During Shoulder Arthroplasty
Brief Title: Benzoyl Peroxide and Electrocautery Skin Incision to Eradicate Cutibacterium Acnes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough funding to conduct the project
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, H. Mike Kim, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2095111
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Prosthetic-joint Infection
Keywords: Shoulder arthroplasty; Prosthetic joint infection; Cutibacterium acnes; Benzoyl peroxide; Electrocautery
MeSH Terms: interventions — Benzoyl Peroxide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Electrocautery-incision alone group (Active Comparator): The skin inicsion will be made using electrocautery during shoulder replacement in patients assigned this group with no other preoperative treatment.
  Interventions: Procedure: Electrocautery surgical skin incision
- Electrocautery-incision and BPO group (Experimental): Patients assigned in this group will undergo an application of topical benzoyl peroxide to the shoulder skin prior to shoulder replacement surgery in addition to their skin incision being made using electrocautery.
  Interventions: Drug: Benzoyl Peroxide Topical; Procedure: Electrocautery surgical skin incision

INTERVENTIONS:
Drug: Benzoyl Peroxide Topical — Topical benzoyl peroxide cream will be applied to the shoulder skin twice a day for 2 days leading up to and in the morning of surgery.
  Arms: Electrocautery-incision and BPO group
Procedure: Electrocautery surgical skin incision — The skin incision will be made entirely using electrocautery at the beginning of shoulder replacement.

SUMMARY:
The goal of this prospective randomized clinical trial is to investigate the potential synergistic effect of combination of topical benzoyl peroxide and making skin incision with electrocautery on preventing surgical wound contamination from Cutibacterium acnes (C. acnes) in patients undergoing shoulder replacement.

The main question it aims to answer is:

• Will the combined use of topical application of benzoyl peroxide and making skin incision using electrocautery decrease the positive culture rates of C. acnes in the surgical field?

Participants will be asked to apply topical benzoyl peroxide to the shoulder skin prior to their shoulder replacement surgery if they are randomized in the treatment group. The skin incision will be made using electrocautery in both the control and treatment groups. Microbiology swab cultures will be taken during shoulder replacement surgery to compare the positive culture rates for C. acnes between the groups.

DETAILED DESCRIPTION:
Periprosthetic joint infection (PJI) following shoulder arthroplasty is not only detrimental to patients but also immensely burdensome on our healthcare system. The rate of PJI following shoulder arthroplasty is estimated between 0.80 and 1.46%, with the incidence expected to increase as shoulder arthroplasty continues to become more common. Cutibacterium acnes (C. acnes), a gram-positive anaerobe commonly found in sebaceous glands, is the most common causative organism behind PJI of shoulder arthroplasty. The human shoulder skin is heavily colonized with C. acnes, and studies showed that the current standard sterilization practices are not able to completely remove C. acnes from the surgical field. It is theorized that when skin incisions are made, the sebaceous glands in the skin are also cut open, releasing C. acnes and contaminating gloves, instruments, and eventually the surgical field during subsequent part of the procedure. Preventing C. acnes contamination could potentially decrease PJI significantly after shoulder arthroplasty.

Electrocautery has been routinely used for tissue dissection and hemostasis. Studies have demonstrated the safety and efficacy of electrocautery for making skin incisions as an alternative to a scalpel blade. It is hypothesized that the high temperatures generated at the tip of an electrocautery electrode might potentially heat up and destroy the exposed C. acnes at the incised dermal edge. This hypothesis has been recently proven in a randomized clinical trial conducted at the investigators' institution. Cultures taken from the incised dermal edge immediately after making skin incision with electrocautery resulted in zero positive C. acnes culture compared to a 31% positive culture rate observed with incisions made with scalpel blades. Although it appeared that electrocautery initially eliminated C. acnes from the incision sites, cultures taken from surgeon's gloves and instruments towards the end of the case were found to be positive for C. acnes. All positive cultures were exclusively from male patients. It remains to be answered whether the benefits of electrocautery are only temporary or if the skin surrounding the incision site remains a source for potential contaminant bacteria that current skin prep methods are unable to address.

Topical benzoyl peroxide (BPO) has been widely used as an agent for acne vulgaris, also caused by the same C. acnes bacterium. Studies have investigated the benefits of topical BPO application before open shoulder procedures in reducing C. acnes colonization at the surgical site skin. Compared to conventional skin prep methods, the addition of BPO was found to be significantly more effective in reducing C. acnes from the skin. Based on this finding, it seems to be an interesting yet logical hypothesis that combining topical BPO with electrocautery skin incision might have a synergistic effect against C. acnes. However, no studies to date have sought to examine this hypothesis. To this end, the investigators propose a prospective randomized clinical trial to test this hypothesis through the following specific aim.

Specific Aim: To investigate whether a topical BPO skin prep combined with electrocautery skin incision will lead to a critical reduction of positive C. acnes culture rates in the surgical field compared to electrocautery skin incision alone in shoulder arthroplasty patients.

Methods: Sixty-four male patients (based on a priori sample size calculation) undergoing primary shoulder arthroplasty will be randomized into 2 groups - electrocautery incision alone vs. electrocautery incision combined with BPO skin prep. The investigators will obtain a swab culture for C. acnes from the incised dermal edge immediately after skin incision, and then toward the end of procedure (immediately before humeral component insertion), the investigators will obtain another set of cultures from the incised dermal edge, surgeon's gloves, and joint synovium. The primary outcome measure will be the positive culture rates for C. acnes compared between the 2 groups.

Hypothesis: Compared to the electrocautery incision alone group, the group that receives electrocautery incision combined with BPO skin prep will yield significantly lower positive culture rates for C. acnes in the samples taken later during the procedure, but not in the samples taken from the dermal edge immediately after skin incision.

Expected outcomes and impact: It is expected that the combination of electrocautery skin incision and BPO will lead to a significant reduction of C. acnes positive culture rates in the surgical field. This study, if supported by the study finding, could potentially help understand the underlying mechanism of unexpected positive C. acnes cultures in shoulder arthroplasty and may provide a cost-effective solution for this common clinical problem.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patients (>18 years old) who will undergo primary shoulder arthroplasty (either anatomic or reverse) secondary to osteoarthritis, cuff tear arthropathy, or massive irreparable rotator cuff tear.

Exclusion Criteria:

* History of ipsilateral open shoulder procedures
* History of ipsilateral shoulder infection (either native or postoperative infection)
* Intake of any preoperative antibiotics within one month prior to index surgery
* Active acne at surgical site
* History of psoriatic or eczematous lesions to the surrounding shoulder region
* History of allergic reactions to benzoyl peroxide
* Planned for revision arthroplasty surgery
* Minors under the age of 18 years old
* Female patients
* Prisoners
* Workers compensation insurance status
* Surgery planned for acute proximal humerus fracture or fracture sequelae (nonunion or malunion)
* Patients who cannot understand English well enough to adequately provide informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Late dermis C. acnes culture rates | Within 14 days of shoulder replacement surgery
  Positive C. acnes culture rates from samples taken from the incised dermis during the later part of shoulder replacement

SECONDARY OUTCOMES:
Mid-procedure synovium C. acnes culture rates | Within 14 days of shoulder replacement surgery
  Positive C. acnes culture rates from samples taken from the synovium during the middle of the shoulder replacement

CONTACTS AND LOCATIONS:
Overall Officials: Hyunmin M Kim, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual patients' deidentified demographic information (age and sex only) and microbiology culture results can be shared with other researchers upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From May 2023 to May 2025